CLINICAL TRIAL: NCT00756444
Title: A Randomized Phase 2 Pharmacokinetic Trial of Chemotherapy With or Without Panitumumab in Patients With Metastatic and/or Recurrent Squamous Cell Carcinoma of the Head and Neck (Amended Version 20-March-2009)
Brief Title: A Randomized Phase 2 Pharmacokinetic Trial of Chemotherapy With or Without Panitumumab in Patients With Metastatic and/or Recurrent Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080008
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: PK Study, Metastatic Recurrent
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence | interventions — Panitumumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Panitumumab plus Chemotherapy (Active Comparator): Subjects receiving cisplatin and 5/FU and receiving Panitumumab who have with Metastatic and/or Recurrent Squamous Cell Carcinoma of the Head and Neck
  Interventions: Drug: Panitumumab
- Chemotherapy Alone (Active Comparator): Subjects receiving cisplatin and 5/FU and not receiving Panitumumab who have with Metastatic and/or Recurrent Squamous Cell Carcinoma of the Head and Neck
  Interventions: Drug: Cisplatin; Drug: 5FU

INTERVENTIONS:
Drug: Panitumumab — This is a PK study comparing Panitumumab plus Chemotherapy to Chemotherapy alone
  Arms: Panitumumab plus Chemotherapy
Drug: Cisplatin — This is a PK study comparing Panitumumab plus Chemotherapy to Chemotherapy alone
  Arms: Chemotherapy Alone
Drug: 5FU — This is a PK study comparing Panitumumab plus Chemotherapy to Chemotherapy alone
  Arms: Chemotherapy Alone

SUMMARY:
Study 20080008 was a PK sub-study to study 20050251[Japan 20050251A]. This PK protocol was amended 20-March-2009 and is now a Phase 2 stand alone study. There are no sites participating in the U.S.

This study is designed to estimate the effect of panitumumab on the PK of cisplatin and 5-FU in subjects receiving cisplatin and 5-FU with or without panitumumab.

To maximize any potential effect of panitumumab on the PK of cisplatin and 5-FU, the collection of PK samples of cisplatin and 5-FU will be taken during cycle 2 of the study, the point at which the PK of panitumumab is expected to be at steady-state after a dose of 9 mg/kg given every 3 weeks.

DETAILED DESCRIPTION:
Study Phase: 2 Indication: Metastatic and/or Recurrent Squamous Cell Carcinoma of the Head and Neck Primary Objective: To estimate the effect of administration of 9 mg/kg Q3W of panitumumab on the area under the curve (AUC) of total plasma cisplatin-derived platinum levels and the average concentration at steady state (Css) of 5-fluorouracil (5-FU) in subjects who are receiving cisplatin and 5-FU.

Secondary Objective(s): To estimate the effect of administration of 9 mg/kg Q3W of panitumumab on the maximum concentration (Cmax) of total plasma cisplatin-derived platinum levels, AUC and Cmax of free plasma cisplatin-derived platinum in subjects who are receiving cisplatin and 5-FU.

Hypotheses: This is an estimation sub-study rather than formal hypothesis testing, the following will be estimated:

1. The effect of administration of 9 mg/kg Q3W of panitumumab at steady state on the pharmacokinetics of cisplatin will be estimated based on the ratio for AUC with:without panitumumab of total plasma cisplatin-derived platinum levels. Total plasma cisplatin-derived platinum levels will be the focus since it has been shown in the literature that there are correlations between total plasma cisplatin-derived platinum levels and nephrotoxicity and tumor response (Desoize et al, 1991).
2. The effect of administration of 9 mg/kg Q3W of panitumumab at steady state on the pharmacokinetics of 5-FU assessed based on the average concentration at steady state (Css) of 5-FU.

Study Design: Study 20080008 is a PK study.

This study is designed to estimate the effect of panitumumab on the PK of cisplatin and 5-FU in subjects receiving cisplatin and 5-FU with or without panitumumab.

To maximize any potential effect of panitumumab on the PK of cisplatin and 5-FU, the collection of PK samples of cisplatin and 5-FU will be taken during cycle 2 of the study, the point at which the PK of panitumumab is expected to be at steady-state after a dose of 9 mg/kg given every 3 weeks.

Primary and Secondary Endpoints: The primary endpoints for this study are the ratio of geometric means (with:without panitumumab) for AUC of total plasma cisplatin-derived platinum and average concentration at steady sate (Css) of 5-FU measured at cycle 2 at which time panitumumab levels are anticipated to be at steady state. Secondary endpoints are the ratio of geometric means (with:without panitumumab) for 1) Cmax of total plasma cisplatin-derived platinum and 2) Cmax and AUC of free plasma cisplatin-derived platinum measured at cycle 2.

Sample Size: Approximately 45 subjects will participate in Study 20080008. At least fifteen evaluable subjects (defined as providing sufficient PK samples to permit calculation of AUC for total plasma cisplatin-derived platinum and average concentration at steady state for 5-FU in cycle 2) per arm will be required. Additional subjects will be sequentially included until at least fifteen evaluable subjects per arm are achieved. It is therefore estimated that approximately 45 subjects will need to participate in the study to obtain 30 evauable subjects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck (SCCHN) or its variants (eg, basaloid squamous cell carcinoma and adenosquamous cell carcinoma) of the oral cavity, oropharynx, hypopharynx, or larynx
* Diagnosis of metastatic disease and/or recurrent disease following locoregional therapy and determined to be incurable by surgery or radiotherapy
* Subjects who have received radiation as primary therapy are eligible if locoregional recurrence is in the field of radiation and has occurred ≥6 months after the completion of radiation therapy. Subjects whose locoregional recurrence is solely outside the field of radiation are eligible if the recurrence has occurred ≥ 3 months after the completion of radiation therapy.
* Measurable or non measurable disease. Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to randomization.
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* Man or woman ≥ 18 years of age
* Hematological function, as follows (≤ 10 days prior to randomization):

Absolute neutrophil count (ANC) ≥1.5 x 109/L Platelet count ≥ 100 x 109/L Hemoglobin ≥ 9 g/dL - Renal function, as follows (≤ 10 days prior to randomization):

Creatinine clearance (CrCl) ≥ 50 mL/min calculated by the Cockcroft Gault method as follows:

Male creatinine clearance = (140 age) x (weight in Kg) / (serum Cr x 72) Female creatinine clearance = (140 age) x (weight in Kg) x 0.85 / (serum Cr x 72)

- Hepatic function, as follows (≤ 10 days prior to randomization): Aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN) (≤ 5 x ULN if liver metastases) Alanine aminotransferase (ALT) ≤ 3 x ULN (≤ 5 x ULN if liver metastases) Total bilirubin ≤ 1.5 x ULN

- Electrolytes, as follows (≤ 10 days prior to randomization): Magnesium ≥ lower limit of normal (LLN)

- Negative pregnancy test ≤ 72 hours prior to randomization (females of childbearing potential only)

Exclusion Criteria:

* Documented or symptomatic central nervous system metastases
* History of another primary cancer, except:

Curatively treated in situ cervical cancer, or Curatively resected non melanoma skin cancer, or Other primary solid tumor curatively treated with no known active disease present and no treatment administered for ≥ 2 years prior to randomization

* Subjects whose only site of metastatic disease is a single spiculated lung nodule are assumed to have a second lung primary and are excluded unless there is unequivocal pathological confirmation of metastasis of the SCCHN primary
* Nasopharyngeal carcinoma
* Prior systemic treatment for metastatic and/or recurrent SCCHN Subjects with recurrent disease may have received re irradiation; however subjects who received chemotherapy concomitantly with re irradiation are excluded
* Prior systemic chemotherapy for SCCHN as part of the initial multimodality treatment for locally advanced disease if completed < 6 months prior to randomization
* Prior cisplatin containing induction chemotherapy followed by cisplatin containing chemoradiotherapy
* Prior anti EGFr antibody therapy (eg, cetuximab) or treatment with small molecule EGFr inhibitors (eg, gefitinib, erlotinib, lapatinib)
* Subjects requiring immunosuppressive agents (eg, methotrexate and cyclosporine), however corticosteroids are allowed
* Known allergy or hypersensitivity to any component of the study drugs
* Major surgery requiring general anesthesia and a significant incision (ie, larger than what is required for placement of central venous access, percutaneous feeding tube, or biopsy) ≤ 28 days or minor surgery (excluding central venous catheter placement, percutaneous feeding tube, and biopsy) ≤ 14 days prior to randomization. Subjects must have recovered from surgery related toxicities.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year prior to randomization
* History of interstitial lung disease eg, pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest computerized tomography (CT) scan
* Symptomatic peripheral neuropathy grade ≥ 2 based on the Common Terminology Criteria for Adverse Events (CTCAE) v3.0
* Grade ≥ 3 hearing loss based on the CTCAE v3.0 Auditory/Ear (Hearing [without monitoring program])
* Subjects not recovered from all previous acute radiotherapy related toxicities
* Active infection requiring systemic treatment or any uncontrolled infection ≤ 14 days prior to randomization
* Known positive test for human immunodeficiency virus (HIV) infection, hepatitis C virus, chronic hepatitis B infection (testing is not required in the absence of clinical suspicion)
* Any co morbid condition that would increase risk of toxicity (eg, suspected or confirmed dihydropyrimidine deficiency)
* Other investigational procedures are excluded
* Subject currently is enrolled in or ≤ 30 days since ending other investigational device or drug study(s), or subject is receiving other investigational agents(s)
* Subject who is pregnant or breast feeding
* Man or woman of child bearing potential not consenting to use adequate contraceptive precautions ie, double barrier contraceptive methods (eg, diaphragm plus condom) during the course of the study and for 6 months after the last investigational product(s) administration for women, and 1 month for men
* Subject unwilling or unable to comply with study requirements
* Previously randomized into this study or Amgen study 20050251
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-10-21 (Actual); Primary Completion 2012-03-30 (Actual); Study Completion 2012-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women ≥ 18 years of age with metastatic and/or recurrent squamous cell carcinoma of the head and neck were enrolled from 21 October 2008 to 23 August 2011. This study was conducted at 15 centers in Argentina, Brazil, France, Japan, Romania, and Russia.
Pre-assignment Details: Patients were screened at 15 sites to determine eligibility. Using an IVRS, eligible subjects were randomized to panitumumab plus cisplatin and 5-FU or cisplatin and 5-FU alone. It was estimated that approximately 45 subjects would be needed to obtain 30 evaluable subjects. More than 45 subjects were needed and 67 total subjects were enrolled.
Groups:
- Panitumumab Plus Chemotherapy: Treatment will be administered in cycles repeated every 21 days. On day 1 of each cycle, panitumumab will be administered intravenously, prior to chemotherapy, at a dose of 9 mg/kg over 1 hour. Cisplatin will be administered intravenously on day 1 at a dose of 100 mg/m2 over 1 hour. 5-FU will be administered at a dose of 1000 mg/m2/day by continuous intravenous infusion on day 1 to 4 (96 hours).
- Chemotherapy Alone: Treatment will be administered in cycles repeated every 21 days. Cisplatin will be administered intravenously on day 1 at a dose of 100 mg/m2 over 1 hour. 5-FU will be administered at a dose of 1000 mg/m2/day by continuous intravenous infusion on day 1 to 4 (96 hours).
Period: Overall Study
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Started | 33 | 34
Completed | 18 | 13
Not Completed | 15 | 21
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 5 | 4
Not completed — Disease Progression | 2 | 7
Not completed — Ineligibility Determined | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (7.5) | 58.3 (9.1) | 57.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Total Plasma Cisplatin-derived Platinum Levels With and Without the Presence of Panitumumab
Description: AUC refers to area under the concentration curve from time 0 to last measurable concentration. AUC of total plasma cisplatin-derived platinum levels is estimated both for subjects receiving cisplatin with panitumumab and for subjects receiving cisplatin without panitumumab.
Time Frame: Levels measured at 0.5, 1, 2, 3, 4, 6 and 24 hours following start of cycle 2 cisplatin infusion
Population: Subjects who receive at least 2 cycles of assigned treatment and who have sufficient plasma collection to derive AUC
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Panitumuab Plus Chemotherapy: Treatment will be administered in cycles repeated every 21 days. On day 1 of each cycle, panitumumab will be administered intravenously, prior to chemotherapy, at a dose of 9 mg/kg over 1 hour. Cisplatin will be administered intravenously on day 1 at a dose of 100 mg/m2 over 1 hour. 5-FU will be administered at a dose of 1000 mg/m2/day by continuous intravenous infusion on day 1 to 4 (96 hours).
Arm/Group | Panitumuab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 23 | 16
ng*hr/mL | 58000 (9530) | 62300 (10200)

2. Primary Outcome: Steady-state Plasma Concentrations (Css) for 5-FU With and Without the Presence of Panitumumab
Description: Steady-state plasma concentrations (Css) of 5-FU were estimated as the mean of two or more evaluable concentrations at 24, 72, and 96 hours after the start of 5-FU infusion. Css is estimated both for subjects receiving 5-FU with panitumumab and for subjects receiving 5-FU without panitumumab
Time Frame: 24 to 96 hours following start of cycle 2 infusion with 5-FU
Population: Subjects who receive at least 2 cycles of assigned treatment and who have sufficient plasma collection to derive Css
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panitumuab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 22 | 13
ng/mL | 328 (180) | 378 (184)

ADVERSE EVENTS:
Time Frame: 54 Weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  Summary of Adverse Events includes only those subjects who received at least one dose of investigational product.
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone | Total
Serious Adverse Events (participants affected / at risk) | 11/33 | 8/34 | 19/67
Other Adverse Events (participants affected / at risk) | 33/33 | 33/34 | 66/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Chemotherapy (N=33) | Chemotherapy Alone (N=34) | Total (N=67)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Performance status decreased (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pharyngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Carotid artery thrombosis (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 2
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chest tube insertion (Surgical and medical procedures) | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Chemotherapy (N=33) | Chemotherapy Alone (N=34) | Total (N=67)
Anaemia (Blood and lymphatic system disorders) | 17 | 16 | 33
Granulocytopenia (Blood and lymphatic system disorders) | 2 | 4 | 6
Leukopenia (Blood and lymphatic system disorders) | 7 | 12 | 19
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 16 | 15 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 10 | 18
Deafness (Ear and labyrinth disorders) | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3
Constipation (Gastrointestinal disorders) | 4 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 10
Nausea (Gastrointestinal disorders) | 17 | 19 | 36
Oral pain (Gastrointestinal disorders) | 2 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 8 | 1 | 9
Vomiting (Gastrointestinal disorders) | 11 | 9 | 20
Asthenia (General disorders) | 11 | 6 | 17
Fatigue (General disorders) | 3 | 0 | 3
Injection site reaction (General disorders) | 2 | 0 | 2
Mucosal inflammation (General disorders) | 2 | 2 | 4
Pyrexia (General disorders) | 4 | 2 | 6
Xerosis (General disorders) | 2 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 2
Paronychia (Infections and infestations) | 5 | 0 | 5
Pneumonia (Infections and infestations) | 0 | 2 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Blood creatinine increased (Investigations) | 4 | 5 | 9
Blood urea increased (Investigations) | 1 | 3 | 4
Creatinine renal clearance decreased (Investigations) | 0 | 4 | 4
Weight decreased (Investigations) | 10 | 10 | 20
Decreased appetite (Metabolism and nutrition disorders) | 9 | 8 | 17
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 0 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 10 | 27
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 | 0 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 0 | 10
Rash (Skin and subcutaneous tissue disorders) | 15 | 0 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.